CLINICAL TRIAL: NCT01107067
Title: Phase IV Study to Investigate the Effect of Testosterone Treatment on Paraoxonase Level in Male Patients With Hypogonadotrophic Hypogonadism
Brief Title: Testosterone Replacement Therapy Decreases Plasma Paraoxonase 1 Enzyme Activity In Male Patients With Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Gulhane School of Medicine Department of Endocrinology and Metabolism, Gulhane School of Medicine Department of Endocrinology and Metabolism
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: aa001
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2008-05

CONDITIONS: Hypogonadism
Keywords: hypogonadism; paraoxonase; Hipogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- testosterone replacement therapy (Experimental)
  Interventions: Drug: Sustanon

INTERVENTIONS:
Drug: Sustanon — 250 mg/21 days
  Other Names: no name

SUMMARY:
The purpose of this study is investigating the effect of testosterone treatment on paraoxonase level in male patients with hypogonadotrophic hypogonadism

ELIGIBILITY:
Inclusion Criteria:

* Volunteers patients with hypogonadism

Exclusion Criteria:

* Coronary heart disease
* Other pituitary/hypothalamic disorders or other non-hypogonadism diseases
* None was receiving vitamins, lipid-lowering drugs, or other medications known to interfere with PON1 activity, lipid profile, or gonadal function

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
paraoxonase level after testosterone treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aydoğan AYDOĞDU, Ankara, Turkey (Türkiye)